CLINICAL TRIAL: NCT04890353
Title: Impact of an Immune Modulator Dimethyl Fumarate on Acute Ischemic Stroke
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The interim analysis of another associated study is not very effective
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: haojunwei4
Record Dates: First submitted 2021-05-11; First posted 2021-05-18 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2021-05

CONDITIONS: Acute Ischemic Stroke
Keywords: Dimethyl Fumarate; acute ischemic stroke; immune modulation
MeSH Terms: conditions — Ischemic Stroke | interventions — Dimethyl Fumarate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard management plus Dimethyl Fumarate (Experimental)
  Interventions: Drug: Dimethyl fumarate
- standard management (No Intervention)

INTERVENTIONS:
Drug: Dimethyl fumarate — Dimethyl fumarate 240mg orally twice daily for 3 consecutive days
  Arms: standard management plus Dimethyl Fumarate

SUMMARY:
The investigators conduct this study to investigate whether oral administration of Dimethyl Fumarate, a Food and Drug Administration-approved drug for multiple sclerosis, is safe and effective in in alleviating neurologic deficits in patients with Acute Ischemic Stroke.

ELIGIBILITY:
Inclusion Criteria:

1. >18 y of age;
2. acute onset of focal neurological deficit consistent with acute ischemic stroke;
3. measurable neurological deficit (NIHSS ≥ 5);
4. anterior-circulation ischemic stroke defined by magnetic resonance angiography (MRA) and Diffusion-Weighted Imaging(DWI);
5. onset of symptom to admission more than 4.5 h and less than 72 h. Patients who arrived within 0-4.5 h poststroke were treated with other medications according to the best accepted medical treatment guidelines.

Exclusion Criteria:

1. Other diseases of the central nervous system
2. There has been neurological disability in the past (mRS score>2)
3. Difficulty swallowing
4. Arrhythmia, atrioventricular block
5. Use of anti-tumor drugs, other immunosuppressive and immunomodulatory drugs
6. Macular edema
7. MRA shows vertebral basilar artery obstruction
8. Hemorrhagic stroke
9. Patients who are known to have hypersensitivity to dimethyl fumarate or any excipients of this product
10. Pregnant and lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) | day 7
  The NIHSS score ranges from 0 to 42 points. The higher the score, the more severe the neurological impairment.
Lesion Volume | day 7
  Measured by MRI.

SECONDARY OUTCOMES:
The Modified Rankin Scale (mRS) | day1
  The mRS score ranges from 0 to 7 points. The higher the score, the more severe the neurological recovery state of stroke patients.
The Modified Rankin Scale (mRS) | day3
  The mRS score ranges from 0 to 7 points. The higher the score, the more severe the neurological recovery state of stroke patients.
The Modified Rankin Scale (mRS) | day7
  The mRS score ranges from 0 to 7 points. The higher the score, the more severe the neurological recovery state of stroke patients.
The Modified Rankin Scale (mRS) | day14
  The mRS score ranges from 0 to 7 points. The higher the score, the more severe the neurological recovery state of stroke patients.
The Modified Rankin Scale (mRS) | day90
  The mRS score ranges from 0 to 7 points. The higher the score, the more severe the neurological recovery state of stroke patients.
National Institutes of Health Stroke Scale (NIHSS) | day 1
  The NIHSS score ranges from 0 to 42 points. The higher the score, the more severe the neurological impairment.
National Institutes of Health Stroke Scale (NIHSS) | day 3
  The NIHSS score ranges from 0 to 42 points. The higher the score, the more severe the neurological impairment.
National Institutes of Health Stroke Scale (NIHSS) | day 14
  The NIHSS score ranges from 0 to 42 points. The higher the score, the more severe the neurological impairment.
National Institutes of Health Stroke Scale (NIHSS) | day 90
  The NIHSS score ranges from 0 to 42 points. The higher the score, the more severe the neurological impairment.
Lesion Volume | day 1
  Measured by MRI.
Lesion Volume | day 3
  Measured by MRI.
Lesion Volume | day 90
  Measured by MRI.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China